CLINICAL TRIAL: NCT04524988
Title: Comparing Surgical Proficiency of Laparoscopic Vaginal Cuff Suturing in Surgically Naïve Learners After Training With Two Different Laparoscopic Simulators: A Randomized Controlled Trial
Brief Title: Comparing Proficiency of Laparoscopic Vaginal Cuff Suturing After Laparoscopic Training in Surgically Naive Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Magdy Milad, MD, Albert B. Gerbie Professor; Chief, Gynecology and Gynecologic Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STU00209340
Record Dates: First submitted 2020-05-17; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Educational Problems

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fundamentals of Laparoscopic Surgery (FLS) (Active Comparator): This group will undergo 2.5h of training on the current standard laparoscopic simulation trainer (FLS), including the following tasks: peg transfer, intracorporeal knot tying and ligating loop.
  Interventions: Procedure: Laparoscopic Simulation Training
- Essentials in Minimally Invasive Gynecology (EMIG) (Experimental): This group will undergo 2.5h of training on a new gynecology-specific laparoscopic simulation trainer (EMIG), including the following tasks: peg transfer, intracorporeal knot tying and running suture.
  Interventions: Procedure: Laparoscopic Simulation Training

INTERVENTIONS:
Procedure: Laparoscopic Simulation Training — All participants underwent 2.5h of training with one of two laparoscopic simulation trainers (FLS or EMIG).

SUMMARY:
Surgically naive premedical and medical students were trained on two different laparoscopic simulation trainers, then tested on the same vaginal cuff suturing model. Video recordings were collected from the vaginal cuff suturing tasks. These recordings were graded by expert gynecologic surgeons using a laparoscopic skills rubric. Their scores were compared to determine if one of the two laparoscopic trainers better prepared surgically naive students to complete a gynecologic surgical task.

DETAILED DESCRIPTION:
Surgically naive premedical and medical students were recruited from June-November 2019. They were block randomized into two laparoscopic simulation training groups: Essentials in Minimally Invasive Gynecology (EMIG) or Fundamentals of Laparoscopic Surgery (FLS). Demographic data was collected from all participants. Participants watched instructional videos specific to their simulation trainer, as well as a video for the vaginal cuff suturing task. Participants then completed a pre-test on a vaginal cuff laparoscopic suturing model. They underwent EMIG or FLS training for approximately 2.5 hours. After training, they completed a post-test on the same vaginal cuff laparoscopic suturing model. Both pre- and post-test tasks were recorded. Video recordings were reviewed and graded by two expert high-volume MIGS surgeons who were masked to participant group (EMIG or FLS) and test phase (pre- or post-test). A modified version of the previously validated GOALS tool was used for grading. Participants also completed a survey rating their confidence level in performing laparoscopic tasks using a 5-point Likert scale after completion of their post-test vaginal cuff suturing task.

ELIGIBILITY:
Inclusion Criteria:

* current student enrolled in premedical internship program at Northwestern during recruitment dates
* current medical student in M1/M2 preclinical years enrolled in accredited medical school
* MD/PhD student in their PhD year(s) enrolled in accredited medical school

Exclusion Criteria:

* medical student in M3/M4 clinical years enrolled in accredited medical school

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Proficiency of surgically naive premedical/medical students at completing a vaginal cuff suturing task following training on one of two laparoscopic simulators | 4 hours
  Using a previously validated laparoscopic skills assessment tool (Global Operative Assessment of Laparoscopic Skills, or GOALS), two expert MIGS surgeons reviewed each video and scored it using a modified version of the GOALS tool. Each participant was ultimately given a GOALS composite score, which was made up of 8 individual skill domains (3 of which were added to make the scoring relevant and specific to the vaginal cuff suturing task). The GOALS scores serve to measure student surgical proficiency at laparoscopic tasks.

SECONDARY OUTCOMES:
Correlation of fine motor skills task experience with laparoscopic surgical task performance | 4 hours
  Demographic data was collected from each participant in a survey prior to their training session. This data included experience with fine motor skills tasks, including video games, sewing and playing an instrument. As above, objective performance scores were obtained after video grading using a modified version of the GOALS tool. GOALS scores from participants with fine motor skills task performance were compared with GOALS scores for participants without the same prior fine motor skills task experience to assess for associations between performance and previous fine motor skill task experience.

OTHER OUTCOMES:
Student-reported confidence on laparoscopic surgical task performance | 4 hours
  All participants completed a survey after training where they rated their confidence in performing individual laparoscopic tasks using a 5-point Likert scale. Scores will be compared between the two study arms to determine if either simulator is associated with higher confidence ratings for completing laparoscopic tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Milad, MD, Principal Investigator — Northwestern University Feinberg School of Medicine; Emily Lin, MD, Study Director — Northwestern University Feinberg School of Medicine
Locations (1):
- 259 E Erie - Northwestern, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No